CLINICAL TRIAL: NCT05035550
Title: Effects of Open-label Placebos Administered Through Telehealth on COVID-related Stress, Anxiety, and Depression
Brief Title: Effects of Open-label Placebos on COVID-related Psychological Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Jason S. Moser, Professor of Psychology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NDP00004435
Record Dates: First submitted 2021-08-12; First posted 2021-09-05 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stress; Anxiety; Depression
Keywords: COVID-19; Non-Deceptive Placebos; Intervention; Telehealth; Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Who Masked: Participant
Masking Description: The control group was blinded to their condition. The intervention group was not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Deceptive Placebo (Experimental): The NDP group was informed that the purpose of the study was to test a mind-body intervention that might help participants deal with the stress and anxiety that they are feeling during the pandemic. The intervention included two videos that introduced the effects of non-deceptive placebos, followed by a presentation on up-to-date non-deceptive placebo research. The participants then received instruction on how they would take their non-deceptive placebos for the next two weeks. Participants were asked to complete daily pill-taking adherence surveys (~5 min) and weekly at midpoint (1-week) and endpoint (2-week).
  Interventions: Behavioral: Non-Deceptive Placebo
- No-Treatment Control (No Intervention): The Control group did not receive an intervention. Instead, participants were informed that the purpose of the study was to track individual psychological and physical health over longer time periods in the context of the pandemic. Participants were asked to complete weekly questionnaires at midpoint (1-week) and endpoint (2-week).

INTERVENTIONS:
Behavioral: Non-Deceptive Placebo — The placebos were ordered through Amazon from Zeebo® (Zeebo, Zeebo Effect, LLC, South Burlington, Vermont, USA). The placebos in this study were blue and white capsules containing Microcrystalline cellulose (an inert fiber). Ingredients include ones that are typically used to make pills including silica, gelatin, titanium dioxide, red #3 food coloring, and blue #1 food coloring. Placebo capsules were free of any active ingredients. These bottles were not branded specifically for the experiment, including the brand name ("Zeebo Relief"), description of the contents, directions, and a disclaimer. The investigators chose to not include a custom label for transparency and in order to increase "non-deceptive" placebo effects. Participants were instructed to take two pills a day, one in the morning and one in the evening.
  Arms: Non-Deceptive Placebo

SUMMARY:
This project aimed to test the efficacy of a telehealth-administered placebo without deception intervention on stress, anxiety, and depression related to the COVID-19 pandemic. Participants were randomized into two groups (open-label placebo vs. no-treatment control). All participants received information on the impact of COVID-19 on psychological health. Participants in the open-label placebo group were instructed to watch an informational video on the beneficial effects of placebos without deception, remotely interact with an experimenter, and take open-label placebo pills twice a day for two weeks. Participants in the no-treatment control group did not receive any intervention. Instead, participants met with an experimenter and reported on their psychological and physical health. The investigators predicted that the placebo without deception group would exhibit substantially reduced stress, depression, and anxiety compared to a no-treatment control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have experienced moderate COVID-19 stress, as assessed by a score of ≥ 35 on the COVID-19 Stress Scale (Taylor et al., 2020).

Exclusion Criteria:

* Non-Michigan residents; self-reported diagnosis of anxiety, depression, ADHD, schizophrenia, bipolar disorder, substance use disorder; currently taking psychotropic medication including antidepressants, anti-anxiety medication or stimulants; allergies or concerns with the placebo pill ingredients; or active diagnosis of COVID-19 at the time of eligibility or enrollment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Moser, Ph.D., Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the IPD used in the analysis for manuscript submission.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be available one year after publication
Access Criteria: IPD will be available upon request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Started | 32 | 32
Completed | 29 | 32
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Deceptive Placebo | No-Treatment Control | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Full Range); unit: years] | 21.22 [18 to 30] | 20.97 [19 to 26] | 21.09 [18 to 30]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 3 | 3 | 6
  Female | 29 | 29 | 58
  Intersex | 0 | 0 | 0
  Not Listed | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American/ American Indian/Alaskan Native/ Indigenous | 0 | 0 | 0
  East Asian (Korean, Japanese, Chinese, etc.) | 0 | 5 | 5
  Southeast Asian (Vietnamese, Cambodian, Filipino, etc.) | 2 | 1 | 3
  South Asian (Indian, Pakistani, Sri Lanka, etc.) | 3 | 3 | 6
  Black/ African American | 0 | 1 | 1
  Latinx/ Hispanic | 0 | 0 | 0
  Middle Eastern/ North African | 0 | 1 | 1
  Native Hawaiian/ Pacific Islander | 0 | 0 | 0
  White/ European | 26 | 18 | 44
  Multiracial | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
COVID Stress Scale (CSS) [Mean (Standard Deviation); unit: units on a scale] — Population: Two participants in the non-deceptive placebo group dropped out before baseline assessment.
  units on a scale
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 34.70 (18.495) | 35.13 (20.500) | 34.92 (19.397)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — Population: Two participants in the non-deceptive placebo group dropped out before baseline assessment.
  units on a scale
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 22.47 (6.632) | 20.34 (7.489) | 21.37 (7.109)
PROMIS Anxiety Short Form [Mean (Standard Deviation); unit: units on a scale] — Population: Two participants in the non-deceptive placebo group dropped out before baseline assessment.
  units on a scale
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 25.77 (6.694) | 23.69 (6.621) | 24.69 (6.684)
Center for Epidemiological Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Population: Two participants in the non-deceptive placebo group dropped out before baseline assessment.
  units on a scale
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 22.80 (10.662) | 20.75 (12.104) | 21.74 (11.383)

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Related Stress
Description: Self-reported COVID-19 related stress was measured using the COVID-19 Stress Scale. The Covid stress scale (CSS) is a 36-item self-report questionnaire that measures stress-related to COVID-19 (Taylor et al., 2020). Participants rated each item on a 0 (not at all) to 4 (extremely) scale. For the purposes of this study, only total scores were calculated. Total score ranges from 0-144 with higher scores indicating greater COVID-related stress.
Time Frame: COVID-19 related stress was measured at Baseline (Day 1), Midpoint (Day 7), and Endpoint (Day 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline (Day 1) | 34.93 (18.78) | 35.13 (20.50)
  Midpoint (Day 7) | 26.24 (17.29) | 32.37 (18.51)
  Endpoint (Day 14) | 12.28 (16.01) | 28.34 (20.61)

2. Primary Outcome: Perceived Stress
Description: Self-reported perceived stress was measured using the Perceived Stress Scale (PSS). The Perceived Stress Scale (PSS) is a 10-item self-report questionnaire that assesses the extent to which different situations affect our perceptions of stress during the last month (Cohen, 1994). The scale was modified for the current study in order to measure ratings of perceived stress over the past 7 days. Participants rated each item on a 0 (never) to 4 (very often) scale. Total score ranges from 0-40 with higher scores indicating greater perceived stress.
Time Frame: Perceived stress measured at Baseline (Day 1), Midpoint (Day 7), and Endpoint (Day 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline (Day 1) | 22.52 (6.74) | 20.34 (7.49)
  Midpoint (Day 7) | 17.24 (7.19) | 17.98 (7.12)
  Endpoint (Day 14) | 15.00 (5.91) | 17.78 (7.12)

3. Primary Outcome: Anxiety
Description: Self-reported anxiety was measured using the PROMIS Emotional Distress - Anxiety - Short Form. The PROMIS Emotional Distress - Anxiety - Short Form is an 8-item self-report questionnaire that assesses anxiety over the past 7 days in adults. Participants rated each item on a 1 (never) to 4 (always) scale. Total score ranges from 8-40 with higher scores indicating greater anxiety.
Time Frame: Anxiety symptom severity was measured at Baseline (Day 1), Midpoint (Day 7), and Endpoint (Day 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline (Day 1) | 25.62 (6.76) | 23.69 (6.62)
  Midpoint (Day 7) | 22.07 (7.93) | 22.19 (7.46)
  Endpoint (Day 14) | 19.00 (6.02) | 21.81 (7.92)

4. Primary Outcome: Depression
Description: Self-reported anxiety was measured using the Center for Epidemiological Studies - Depression (CES-D) Scale. The Center for Epidemiological Studies - Depression (CES-D) Scale is a 20-item self-report questionnaire that assesses depressive symptoms over the past 7 days. Participants rated each item on a 0 [rarely or none at the time (less than one day)] to 3 [most or all of the time (5 to 7 days)] scale. Total score ranges from 0-60 with higher scores indicating higher levels of depression.
Time Frame: Depression symptom severity was measured at Baseline (Day 1), Midpoint (Day 7), and Endpoint (Day 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline (Day 1) | 22.69 (10.83) | 20.75 (12.10)
  Midpoint (Day 7) | 17.90 (10.26) | 20.76 (12.35)
  Endpoint (Day 14) | 12.93 (8.56) | 18.31 (11.86)

5. Secondary Outcome: Treatment Expectations
Description: Participants in the open-label placebo group rated their expectations of the open-label placebo treatment using representative questions (10-items) from each sub-scale of the Treatment Expectations Questionnaire (TEX-Q; Alberts et al. (2020). Two subscales were calculated from exploratory factor analysis: Expected benefits and Expected harm. The range for expected benefits ranged from 0-10 with higher scores indicating greater benefits from the OLP. The range for expected harm also ranged from 0-10 with higher scores indicating expecting more harm.
Time Frame: Treatment expectations were measured during the administration of the intervention (Day 1) and at the end of the study (Day 14)
Population: Participants in the No-Treatment Control group were not administered the Treatment Expectations Questionnaire because they did not receive any treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 0
score on a scale
  Expected Benefits (Day 1) | 6.30 (2.09) |
  Expected Benefits (Day 14) | 5.21 (2.17) |
  Expected Harm (Day 1) | .53 (1.06) |
  Expected Harm (Day 14) | .32 (.58) |

6. Secondary Outcome: Treatment Adherence
Description: Participants in the open-label placebo group were instructed to take two placebo pills a day for 14 days (28 placebo pills). Treatment adherence was measured as the percentage of placebo pills taken by each participant (number of pills taken / 28 * 100).
Time Frame: Treatment adherence was measured daily for 14 days beginning after intervention administration (Day 1).
Population: Treatment adherence was not measured in the No-Treatment Control group because they did not receive the treatment.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 0
percentage of pills taken | 92.5 (9.7) |

7. Secondary Outcome: Intervention Feasibility
Description: Intervention feasibility was measured using the Feasibility of Intervention Measure (FIM; Weiner et al., 2017). The FIM is a 4-item self-report measure that assesses the extent to which an intervention can be successfully implemented within a given setting. The items are averaged with scores ranging from 1-5 with higher numbers indicating that the OLP intervention is easy to use and doable.
Time Frame: Ratings of intervention feasibility were measured at Endpoint (Day 14)
Population: Intervention feasibility was not measured in the No-Treatment Control group because they did not receive the treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 0
score on a scale | 4.31 (.54) |

8. Secondary Outcome: Intervention Acceptability
Description: Intervention acceptability was measured using the Acceptability of Intervention Measure (AIM; Weiner et al., 2017). The AIM is a 4-item self-report measure that assesses the extent to which an intervention is perceived to be satisfactory, adequate, and appealing. The items are averaged with scores ranging from 1-5 with higher numbers indicating that the OLP intervention is satisfactory and appealing.
Time Frame: Ratings of intervention acceptability were measured at Endpoint (Day 14)
Population: Intervention acceptability was not measured in the No-Treatment Control group because they did not receive the treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 0
score on a scale | 4.03 (.72) |

9. Secondary Outcome: Intervention Appropriateness
Description: Intervention appropriateness was measured using the Intervention Appropriateness Measure (IAM; Weiner et al., 2017). The IAM is a 4-item self-report measure that assesses the extent to which an intervention is perceived to be fitting, relevant, and compatible with a population or setting to address a particular problem. The items are averaged with scores ranging from 1-5 with higher numbers indicating that the OLP intervention is perceived to be fitting, relevant, and compatible with a population or setting to address a particular problem.
Time Frame: Ratings of intervention appropriateness were measured at Endpoint (Day 14)
Population: Intervention Appropriateness was not measured in the No-Treatment Control group because they did not receive the treatment.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
Number analyzed (Participants) | 29 | 0
score on scale | 3.98 (.69) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of the study from February 4, 2021, to May 5, 2021. Each participant was monitored through the study completion, on average of 15 days.
Description: The participants were asked to inform us openly if they were experiencing any adverse events due to the intervention or participation in the study. They were asked at each zoom interaction and asked to contact us in between Zoom sessions.
Arm/Group | Non-Deceptive Placebo | No-Treatment Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT05035550/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT05035550/SAP_001.pdf